CLINICAL TRIAL: NCT02288039
Title: A Pilot Study to Assess the Feasibility and Efficacy of a Social Identity Theory Based Intervention to Improve the Quality of Life of Patients Attending Pulmonary Rehabilitation.
Brief Title: Quality of Life in Pulmonary Rehabilitation: A Social Identity Based Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: Edge Hill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1132
Record Dates: First submitted 2014-10-31; First posted 2014-11-11 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social Identity Goal-Based Intervention (Experimental): Participants will receive collaborative goal-setting
  Interventions: Other: Social Identity goal-based Intervention
- Standard Care (No Intervention): Participants will receive usual standard treatment

INTERVENTIONS:
Other: Social Identity goal-based Intervention — Phase 1: collaborative group discussion in order to establish what group members want to achieve by the end of their 8-week pulmonary rehabilitation programme. Phase 2: further collaborative group discussion with the emphasis on evaluating, monitoring, and providing feedback on goal attainment. Phase 3: focus group interviews with an emphasis on reviewing the goal setting process that patients have engaged with.
  Arms: Social Identity Goal-Based Intervention

SUMMARY:
The main aim of pulmonary rehabilitation is to improve the quality of life of patients that have been diagnosed with chronic lung disease. The challenge for pulmonary rehabilitation is that many patients do not complete their agreed or prescribed training targets which may be related to the way pulmonary rehabilitation is delivered. There is a belief among doctors and other healthcare professionals delivering pulmonary rehabilitation care that patients who are working together as part of a group may better accomplish their agreed training targets (intervention). The intervention aims to encourage members of the group to interact and support each other during the rehabilitation sessions in order to attain agreed pulmonary rehabilitation goals

DETAILED DESCRIPTION:
Previous research indicates that self-management interventions vary, comprising of patient education, action planning, goal setting, cognitive behavioural therapy and motivational interviewing. The delivery of these interventions was largely conducted through individual sessions either face-to-face or telephone conversations, or through the individual distribution of booklet information. As such, research has heavily focused on individual-focused self-management interventions in order to facilitate QoL in COPD patients. It is not surprising that interventions have largely taken an individualistic approach given that sufferers of COPD are diagnosed and treated as individuals (e.g., in hospital, or when visiting the doctor). However, at times COPD management is delivered in groups (e.g., exercise/ education rehabilitation sessions). Indeed, the group-management of COPD treatment for improving the QoL of COPD patients has largely remained unexplored. Therefore, a significant limitation of self-management approaches used to-date concerns the lack of consideration given to group-management interventions. The proposed study therefore aims to address this limitation by investigating the a group-based psychological intervention.

Participants will be assigned to one of two groups: 1) the control group containing standard care; and 2) the intervention group containing standard care plus the intervention. Participants will attend weekly rehabilitation classes for 8 weeks, regardless of the rehabilitation group assigned. In addition, participants will complete a quality of life questionnaire that will ask questions about subjective feelings. The questionnaire will take about 20 minutes to complete. The questionnaire will be completed at the start of the 8-week rehabilitation programme, at the mid-point, and at the end of the rehabilitation programme.

In the intervention arm of the study participants will take part in three focus group discussions. The focus group discussions will be with members of the research team and the rest of your rehabilitation group. The first two sessions help participants plan strategies in order to get the most benefit from the rehabilitation programme. The third session will entail some reflection regarding how well participants thought the programme had addressed their rehabilitation needs. Finally, all participants will complete the quality of life questionnaire again at 3 months after completing the 8-week rehabilitation programme by return stamp-addressed envelope.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are that patients score between 1 and 4 on the Modified Medical Research Council Dyspnoea Scale and have not previously been enrolled on a pulmonary rehabilitation programme

Exclusion Criteria:

* Patients excluded from the study based on these criteria will be assigned to a rehabilitation group not involved in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in Health-related Quality of Life (QoL) scores from baseline | Baseline, 4 weeks, 8 weeks, 12 weeks
  QoL measured using Euroquol EQ-5D-3L and 5L questionnaires

SECONDARY OUTCOMES:
Change in magnitude of social identification score measured using a standardised scale from baseline | Baseline, 4 weeks, 8 weeks, 12 weeks
  The intervention fidelity will be assessed through determining whether social identification has been achieved. This will be measured with four items (from Doosje, Ellemers, & Spears, 1995; e.g. 'Do you see yourself as part of the [COPD exercise group]', 'Are you pleased to be part of the [COPD group]', 'Do you feel strong ties with others in the [COPD exercise group]?', 'Do you identify with others in the [COPD exercise group]. These scales are widely used and amended in this form and are generally found to provide a good index of the theoretical construct of social identification (e.g. see Haslam et al., 2004).
Change in disease-specific quality of life (QoL) scores from baseline | Baseline, 4 weeks, 8 weeks, 12 weeks
  This will be determined using the Chronic Respiratory Questionnaire and the St George's Respiratory Questionnaires. Additionally, the Survey Short Form (SF-36) will also be administered

OTHER OUTCOMES:
Change in anxiety and depression scores from baseline | Baseline, 4 weeks, 8 weeks, 12 weeks
  These will be determined using the Hospital and Anxiety and Depression Scale questionnaire
Change in exercise adherence rates from baseline | Baseline, 4 weeks, 8 weeks
  This is defined as the number of prescribed exercise sessions performed
Change in functional capacity score from baseline | Baseline, 4 weeks, 8 weeks
  This is defined as total distance covered in a 6 minutes walk test.
Healthcare resources use | 12 weeks
  We will assess the use of healthcare resources. We will specifically examine the issue of staff time in association with the delivery of the social identity intervention.
Cost-effectiveness | 12 weeks
  and conduct a cost-effectiveness analysis. We will assess the incremental costs per QALY both from the NHS and societal perspectives.

CONTACTS AND LOCATIONS:
Overall Officials: Bashir Matata, PhD, Study Director — Liverpool Heart & Chest Hospital
Locations (1):
- Liverpool Heart & Chest Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iyer A, Jetten J, Tsivrikos D, Postmes T, Haslam SA. The more (and the more compatible) the merrier: multiple group memberships and identity compatibility as predictors of adjustment after life transitions. Br J Soc Psychol. 2009 Dec;48(Pt 4):707-33. doi: 10.1348/014466608X397628. Epub 2009 Feb 5. PMID 19200408
- [Background] Haslam SA, O'Brien A, Jetten J, Vormedal K, Penna S. Taking the strain: social identity, social support, and the experience of stress. Br J Soc Psychol. 2005 Sep;44(Pt 3):355-70. doi: 10.1348/014466605X37468. PMID 16238844
- [Background] Veenstra K, Haslam SA, Reynolds KJ. The psychology of casualization: evidence for the mediating roles of security, status and social identification. Br J Soc Psychol. 2004 Dec;43(Pt 4):499-514. doi: 10.1348/0144666042565380. PMID 15601506
- [Derived] Levy AR, Matata B, Pilsworth S, Mcgonigle A, Wigelsworth L, Jones L, Pott N, Bettany M, Midgley AW. An intervention for pulmonary rehabilitators to develop a social identity for patients attending exercise rehabilitation: a feasibility and pilot randomised control trial protocol. Pilot Feasibility Stud. 2018 Jan 27;4:40. doi: 10.1186/s40814-018-0238-z. eCollection 2018. PMID 29423258